CLINICAL TRIAL: NCT02807740
Title: To Rehabilitate With Virtual Reality: To Evaluate the Effect of Virtual Reality on Cardiocirculatory System and on Balance in a Sample of Healthy Subject and Patients Affected by Parkinson Disease
Brief Title: Virtual Reality in Parkinson Disease
Acronym: VRPark
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Costanza Pazzaglia, Researcher, Fondazione Don Carlo Gnocchi Onlus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Prot. n.5/2016/CE_FdG/SA
Record Dates: First submitted 2016-05-31; First posted 2016-06-21 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Parkinson Disease
Keywords: Virtual Reality; Rehabilitation; Cardiocirculatory system; Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Virtual Reality (Experimental): Patients will be treated with a virtual reality rehabilitation program
  Interventions: Other: Virtual reality
- Conventional Rehabilitation Program (Other): Patients will be treated with a conventional rehabilitation program.
  Interventions: Other: Conventional rehabilitation program

INTERVENTIONS:
Other: Virtual reality — Each session will consist of multiple exercises. These ones are already described, each exercise will be performed by the patient for 4 minutes followed by a 1 minute of rest.
  Other Names: VR rehabilitation group
  Arms: Virtual Reality
Other: Conventional rehabilitation program — In each C rehabilitation session, patients underwent 3 phases: 1) Warm-up phase: passive mobilization of main joints and muscular strengthen of lower limbs; 2) Active phase (both standing than seated): exercises of motor coordination with upper and lower limbs, balance training, start and stop exercises, deambulation training; 3) cool-down phase (with seated patient): manipulation exercises, mobilization exercises, respiratory exercises.
  Other Names: C rehabilitation group
  Arms: Conventional Rehabilitation Program

SUMMARY:
Patients affected by Parkinson disease (PD) can benefit from rehabilitation although the evidences are scattered. In the last years there are increased evidences that virtual reality can improve functional outcome in Parkinson's disease. No evidences are known concerning the cardiological safety and effect on balance of Virtual Reality. The aim of this study is to compare a virtual reality rehabilitation program versus a conventional one in a sample of patients affected by mild to moderate Parkinson and to collect data on cardiological effects.

DETAILED DESCRIPTION:
This study will be a prospective, single-blinded, randomized controlled trial aimed to compare two different rehabilitation programs in PD disease and to evaluate the effect of Virtual Reality on cardiocirculatory system.

Patients will undergo Conventional or Virtual Reality Rehabilitation Program for 6 consecutive weeks, 3-times in a week for a 40 minute session. Moreover, in order to acquire data on cardiocirculatory system during the first and the last sessions an Holter- electrocardiography will be used. Data will be compared with healthy subjects (matched for age and gender).

The used protocols are reported below.

Conventional (C) Rehabilitation Program The Conventional rehabilitation program will be performed according to the " Royal Dutch Society for Physical Therapy Guidelines for physical therapy in patients with Parkinson's disease". In each C rehabilitation session, patients will undergo 3 phases: 1) Warm-up phase: passive mobilization of main joints and muscular strengthen of lower limbs; 2) Active phase (both standing than seated): exercises of motor coordination with upper and lower limbs, balance training, start and stop exercises, deambulation training; 3) cool-down phase (with seated patient): manipulation exercises, mobilization exercises, respiratory exercises.

Virtual Reality (VR) Rehabilitation Program Each session will consist of multiple exercises. These ones are described below, each exercise will be performed by the patient for 4 minutes followed by a 1 minute of rest.

Exercise 1 (named Trumpet H2D1): patients placed in the center of the room and asked to randomly touch a moving trumpet displayed on the wall screen. When the trumpet will be reached by patient's arm, it will disappear giving out a sound.

Exercise 2 (named Pink rose hemiarch left and right H1D2): patients placed in the center of the room and asked to touch the rose projected on the wall screen as a hemiarch, in this exercise the sequence of rose to touch and therefore the distance between the target and the patient will be decided by the physical therapist.

Exercise 3 (named Doggy): patients placed in the center of the room and asked to lead a dog in the four corner of the wall screen. Patients will be free to move in the room.

Exercise 4 (named Eggs): patients placed in the center of the room and asked to touch as fast as possible eggs projected in the wall screen in a random order. When the egg will be reached by patient's arm, it will disappear giving out a sound.

Exercise 5 (named Mole): patients placed in the center of the room and asked to reach a mole that will go out from a hole. The patients will know where the mole will be and they will move in the room. When the mole will be reached by patient's arm, it will disappear giving out a sound.

Exercise 6 (named Stay Or Move In Between): patients placed in the center of the room and wre asked to perform the motor task as indicated by physical therapist while maintaining balance between two lateral bars in order not to touch them and not make them sound.

Exercise 7 (named Leaves): patients placed in the center of the room and asked to clean from wall screen as fast as possible all the leaves projected in the wall.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by mild to moderate PD, according to motor examination section (Part III) of the Unified Parkinson's Disease Rating Scale (UPDRS III)
* ability to independently perform motor rehabilitation
* absence of cognitive impairment (MMSE >25)

Exclusion Criteria:

* severe hearing loss and/or visual deficit
* serious comorbidity making impossible to perform rehabilitation (postural hypotension, heart disease, stroke, severe shoulder-hip disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-05; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Balance Berg Scale (BBS) | Patients will be evaluated at baseline (T0) and at the end of each rehabilitation program (T1), lasting 6 weeks
  It is a 14-item scale that rates each function from 0 (worst) to 4 (best) along a dependence-independence continuum. This summative scale measures balance abilities seen during tasks involving sitting, standing, and positional changes. Total scores are indicative of overall balance abilities, with scores interpreted in the following manner: 0 to 20, wheelchair bound; 21 to 40, walking with assistance; and 41 to 56, independent.This scale has been previously validated in PD patients

SECONDARY OUTCOMES:
Change from Baseline Dynamic gait index (DGI) | Patients will be evaluated at baseline (T0) and at the end of each rehabilitation program (T1), lasting 6 weeks
  is an outcome measure used to characterize mobility performance, specifically the ability to adapt gait to complex walking tasks associated with walking in community environments. The index has 8 items, the results are reported in a four-point ordinal scale, ranging from 0-3. "0" indicates the lowest level of function and "3" the highest level of function. The total score is 24. A result less than 19/24 is predictive of falls in the elderly, while a result more than 22/24 means safe ambulation.
Change from Baseline Disabilities of the arm, shoulder and hand scale (DASH) | Patients will be evaluated at baseline (T0) and at the end of each rehabilitation program (T1), lasting 6 weeks
  is a 30-item, self-report questionnaire designed to measure physical function and symptoms in people with any of several musculoskeletal disorders of the upper limb. The higher the score, the higher the function.

CONTACTS AND LOCATIONS:
Overall Officials: Isabella Imbimbo, MPC, Study Chair — Fondazione Don Carlo Gnocchi
Locations (1):
- Don Carlo Gnocchi Foundation, Rome, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abbruzzese G, Marchese R, Avanzino L, Pelosin E. Rehabilitation for Parkinson's disease: Current outlook and future challenges. Parkinsonism Relat Disord. 2016 Jan;22 Suppl 1:S60-4. doi: 10.1016/j.parkreldis.2015.09.005. Epub 2015 Sep 3. PMID 26360239
- [Result] Mirelman A, Maidan I, Deutsch JE. Virtual reality and motor imagery: promising tools for assessment and therapy in Parkinson's disease. Mov Disord. 2013 Sep 15;28(11):1597-608. doi: 10.1002/mds.25670. PMID 24132848
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886
- [Derived] Pazzaglia C, Imbimbo I, Tranchita E, Minganti C, Ricciardi D, Lo Monaco R, Parisi A, Padua L. Comparison of virtual reality rehabilitation and conventional rehabilitation in Parkinson's disease: a randomised controlled trial. Physiotherapy. 2020 Mar;106:36-42. doi: 10.1016/j.physio.2019.12.007. Epub 2019 Dec 23. PMID 32026844